CLINICAL TRIAL: NCT03480503
Title: Serum apelin12 in Acne Vulgaris
Brief Title: Apelin12 in Acne Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Abdelaziz, Principal Investigator, Assiut University
Other Study IDs: SAAA
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acne Vulgaris
Keywords: Apelin12
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The venous blood sample will be taken from acne patients and control group after fasting for 10-12 hours and the following will be done:
  Fasting blood glucose. Complete lipid profile. Serum level of apelin-12 will be measured using enzyme linked immunosorbent assay(ELISA) technique .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Patients with acne vulgaris , measurement of serum apelin12 by using ELISA technique ,complete lipid profile and fasting blood glucose.
- Control group: Healthy control volunteers, measurement of serum apelin12 by using ELISA technique ,complete lipid profile and fasting blood glucose.

SUMMARY:
Acne vulgaris is a common chronic inflammatory disease of the pilosebaceous unit which is characterized by the formation of non-inflammatory open and closed comedones and inflammatory papules, pustules, nodules and cysts.

It is a multifactorial disease that affects mostly adolescent population. Acne appears very early in puberty during the preteen years, often before menarche in girls. Because many adolescents have acne, it is difficult to predict which individuals are prone to severe cases.

The pathogenesis of acne is complex, with strong evidence supporting the involvement of follicular hyperkeratinization, hyperactivity of the sebaceous glands, colonization of Propionibacterium acnes and yeast, and inflammation. Although the importance of androgens in the pathophysiology of acne has been supported by both clinical studies and experimental data, the research evaluating adipokines are very few in patients with acne vulgaris.

DETAILED DESCRIPTION:
Acne lesions may vary in number during the natural course of the disease and multiple measurements have been developed which is based on clinical examination and photographic documentation, to measure the clinical severity.

The Grading of acne based on the type of lesions, affected surface area and their severity that can help in deciding which therapies are needed in each individual. However, no grading system has been accepted universally. The Global Acne Grading System is a quantitative scoring system to assess the severity of acne. According to this score acne was graded as mild, moderate, severe and very severe.

The severity of acne was also graded using the Comprehensive Acne Severity Scale.

Adipokines are proteins that are synthesized and secreted primarily by adipocytes in response to various stimuli, include interleukin 6 and other small molecular weight bioactive proteins such as adiponectin, resistin, leptin, serpin E1 [also known as plasminogen activator inhibitor 1 and endothelial plasminogen activator inhibitor], visfatin (also known as nicotinamide phosphoribosyltransferase), apelin, chemerin, retinol binding protein 4, and monocyte chemoattractant protein 1.

Due to their different biological properties and diverse cellular targets adipokines are involved in a wide array of (patho)physiological processes and are responsible for mediating the inflammatory effects of the adipose tissue in the local tissue environment as well as to different organs via circulation. By detecting alterations in their serum levels also in dermatological diseases such as acne vulgaris and psoriasis, extensive studies have also started in dermatological research to identify the possible targets and the cutaneous sources of these proteins.

Apelin is an endogenous ligand of the previously discovered "orphan" receptor named APJ, isolated from bovine stomach extracts.

It is a product of apelin gene that is located on chromosome Xq25-26.1 and translated as a 77 amino acid prepropeptide. It is processed into several active molecular forms with different biological activities. Apelin belongs to adipokines group because its m-RNA expression has been demonstrated in mature adipocytes in rodents and humans.

Apelin peptide expression has been also demonstrated in several tissues and seems to have different regulatory functions, depending on the expressing tissue, the apelinergic system distribution over such a variety of tissues has suggested that it might play relevant roles in human physiology.

Apelin has been reported to have an effect on appetite, drinking behavior, angiogenesis, and the cardiovascular system. It is regulated by insulin. Apelin might be a novel target for preventing obesity and obesity-related diseases via enhancement of vascular integrity.

Several active apelin forms exist such as apelin-36, apelin-17, apelin-13, and apelin-12.

Apelin-12 is a 12-amino peptide fragment that has been implicated in reducing blood pressure via a nitric oxide mechanism, and is involved in feeding mechanisms via stimulation of cholecystokinin secretion.

It is considered to be one of the most potent isoform of apelin.

The studies evaluating the role of adipokines are very few in patient with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris patients from different ages and sex.

Exclusion Criteria:

* Pregnant and lactating females.
* Local cutaneous infection or any other dermatological diseases.
* Diabetic patients or severe systemic disease such as liver and renal failure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be performed at Department of Dermatology, Venereology and Andrology in Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
serum apelin12 | 12 hour
  blood samples will be taken then measurement of serum apelin12 by using ELISA technique after fasting 12 hours.

SECONDARY OUTCOMES:
Complete lipid profile. | 12hour
  blood samples will be taken and complete lipid profile will be measured after fasting 12 hours by biochemical measurement.
Fasting blood glucose | 7hours
  blood samples will be taken and fasting blood glucose level will be measured after fasting 7 hours by biochemical measurement method.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boucher J, Masri B, Daviaud D, Gesta S, Guigne C, Mazzucotelli A, Castan-Laurell I, Tack I, Knibiehler B, Carpene C, Audigier Y, Saulnier-Blache JS, Valet P. Apelin, a newly identified adipokine up-regulated by insulin and obesity. Endocrinology. 2005 Apr;146(4):1764-71. doi: 10.1210/en.2004-1427. Epub 2005 Jan 27. PMID 15677759
- [Background] Carpene C, Dray C, Attane C, Valet P, Portillo MP, Churruca I, Milagro FI, Castan-Laurell I. Expanding role for the apelin/APJ system in physiopathology. J Physiol Biochem. 2007 Dec;63(4):359-73. PMID 18457011
- [Background] Cordain L, Lindeberg S, Hurtado M, Hill K, Eaton SB, Brand-Miller J. Acne vulgaris: a disease of Western civilization. Arch Dermatol. 2002 Dec;138(12):1584-90. doi: 10.1001/archderm.138.12.1584. PMID 12472346
- [Background] Cox CM, D'Agostino SL, Miller MK, Heimark RL, Krieg PA. Apelin, the ligand for the endothelial G-protein-coupled receptor, APJ, is a potent angiogenic factor required for normal vascular development of the frog embryo. Dev Biol. 2006 Aug 1;296(1):177-89. doi: 10.1016/j.ydbio.2006.04.452. Epub 2006 Apr 27. PMID 16750822
- [Background] De Falco M, De Luca L, Onori N, Cavallotti I, Artigiano F, Esposito V, De Luca B, Laforgia V, Groeger AM, De Luca A. Apelin expression in normal human tissues. In Vivo. 2002 Sep-Oct;16(5):333-6. PMID 12494873
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Farkasfalvi K, Stagg MA, Coppen SR, Siedlecka U, Lee J, Soppa GK, Marczin N, Szokodi I, Yacoub MH, Terracciano CM. Direct effects of apelin on cardiomyocyte contractility and electrophysiology. Biochem Biophys Res Commun. 2007 Jun 15;357(4):889-95. doi: 10.1016/j.bbrc.2007.04.017. Epub 2007 Apr 12. PMID 17466269
- [Background] Gerdes S, Rostami-Yazdi M, Mrowietz U. Adipokines and psoriasis. Exp Dermatol. 2011 Feb;20(2):81-7. doi: 10.1111/j.1600-0625.2010.01210.x. PMID 21255085
- [Background] Kawamata Y, Habata Y, Fukusumi S, Hosoya M, Fujii R, Hinuma S, Nishizawa N, Kitada C, Onda H, Nishimura O, Fujino M. Molecular properties of apelin: tissue distribution and receptor binding. Biochim Biophys Acta. 2001 Apr 23;1538(2-3):162-71. doi: 10.1016/s0167-4889(00)00143-9. PMID 11336787
- [Background] Kitabchi AE, Imseis RE, Bush AJ, Williams-Cleaves B, Pourmotabbed G. Racial differences in the correlation between gonadal androgens and serum insulin levels. Diabetes Care. 1999 Sep;22(9):1524-9. doi: 10.2337/diacare.22.9.1524. PMID 10480520
- [Background] Lee DK, Cheng R, Nguyen T, Fan T, Kariyawasam AP, Liu Y, Osmond DH, George SR, O'Dowd BF. Characterization of apelin, the ligand for the APJ receptor. J Neurochem. 2000 Jan;74(1):34-41. doi: 10.1046/j.1471-4159.2000.0740034.x. PMID 10617103
- [Background] Lehmann HP, Robinson KA, Andrews JS, Holloway V, Goodman SN. Acne therapy: a methodologic review. J Am Acad Dermatol. 2002 Aug;47(2):231-40. doi: 10.1067/mjd.2002.120912. PMID 12140469
- [Background] Liang T, Hoyer S, Yu R, Soltani K, Lorincz AL, Hiipakka RA, Liao S. Immunocytochemical localization of androgen receptors in human skin using monoclonal antibodies against the androgen receptor. J Invest Dermatol. 1993 May;100(5):663-6. doi: 10.1111/1523-1747.ep12472330. PMID 7684056
- [Background] Mesmin C, Fenaille F, Becher F, Tabet JC, Ezan E. Identification and characterization of apelin peptides in bovine colostrum and milk by liquid chromatography-mass spectrometry. J Proteome Res. 2011 Nov 4;10(11):5222-31. doi: 10.1021/pr200725x. Epub 2011 Oct 13. PMID 21939284
- [Background] Najafipour H, Soltani Hekmat A, Nekooian AA, Esmaeili-Mahani S. Apelin receptor expression in ischemic and non- ischemic kidneys and cardiovascular responses to apelin in chronic two-kidney-one-clip hypertension in rats. Regul Pept. 2012 Oct 10;178(1-3):43-50. doi: 10.1016/j.regpep.2012.06.006. Epub 2012 Jul 14. PMID 22796316
- [Background] Ohno S, Yakabi K, Ro S, Ochiai M, Onouchi T, Sakurada T, Takabayashi H, Ishida S, Takayama K. Apelin-12 stimulates acid secretion through an increase of histamine release in rat stomachs. Regul Pept. 2012 Feb 10;174(1-3):71-8. doi: 10.1016/j.regpep.2011.12.002. Epub 2011 Dec 28. PMID 22209991
- [Background] Ozuguz P, Kacar SD, Asik G, Ozuguz U, Karatas S. Evaluation of leptin, adiponectin, and ghrelin levels in patients with acne vulgaris. Hum Exp Toxicol. 2017 Jan;36(1):3-7. doi: 10.1177/0960327116630355. Epub 2016 Jul 11. PMID 26860691
- [Background] Sawane M, Kajiya K, Kidoya H, Takagi M, Muramatsu F, Takakura N. Apelin inhibits diet-induced obesity by enhancing lymphatic and blood vessel integrity. Diabetes. 2013 Jun;62(6):1970-80. doi: 10.2337/db12-0604. Epub 2013 Feb 1. PMID 23378608
- [Background] Seleit I, Bakry OA, Abdou AG, Hashim A. Body mass index, selected dietary factors, and acne severity: are they related to in situ expression of insulin-like growth factor-1? Anal Quant Cytopathol Histpathol. 2014 Oct;36(5):267-78. PMID 25803999
- [Background] Strauss JS, Krowchuk DP, Leyden JJ, Lucky AW, Shalita AR, Siegfried EC, Thiboutot DM, Van Voorhees AS, Beutner KA, Sieck CK, Bhushan R; American Academy of Dermatology/American Academy of Dermatology Association. Guidelines of care for acne vulgaris management. J Am Acad Dermatol. 2007 Apr;56(4):651-63. doi: 10.1016/j.jaad.2006.08.048. Epub 2007 Feb 5. PMID 17276540
- [Background] Sunter D, Hewson AK, Dickson SL. Intracerebroventricular injection of apelin-13 reduces food intake in the rat. Neurosci Lett. 2003 Dec 15;353(1):1-4. doi: 10.1016/s0304-3940(03)00351-3. PMID 14642423
- [Background] Tatemoto K, Hosoya M, Habata Y, Fujii R, Kakegawa T, Zou MX, Kawamata Y, Fukusumi S, Hinuma S, Kitada C, Kurokawa T, Onda H, Fujino M. Isolation and characterization of a novel endogenous peptide ligand for the human APJ receptor. Biochem Biophys Res Commun. 1998 Oct 20;251(2):471-6. doi: 10.1006/bbrc.1998.9489. PMID 9792798
- [Background] Tatemoto K, Takayama K, Zou MX, Kumaki I, Zhang W, Kumano K, Fujimiya M. The novel peptide apelin lowers blood pressure via a nitric oxide-dependent mechanism. Regul Pept. 2001 Jun 15;99(2-3):87-92. doi: 10.1016/s0167-0115(01)00236-1. PMID 11384769
- [Background] Thiboutot D, Gollnick H, Bettoli V, Dreno B, Kang S, Leyden JJ, Shalita AR, Lozada VT, Berson D, Finlay A, Goh CL, Herane MI, Kaminsky A, Kubba R, Layton A, Miyachi Y, Perez M, Martin JP, Ramos-E-Silva M, See JA, Shear N, Wolf J Jr; Global Alliance to Improve Outcomes in Acne. New insights into the management of acne: an update from the Global Alliance to Improve Outcomes in Acne group. J Am Acad Dermatol. 2009 May;60(5 Suppl):S1-50. doi: 10.1016/j.jaad.2009.01.019. PMID 19376456
- [Background] Trayhurn P, Wang B, Wood IS. Hypoxia in adipose tissue: a basis for the dysregulation of tissue function in obesity? Br J Nutr. 2008 Aug;100(2):227-35. doi: 10.1017/S0007114508971282. Epub 2008 Apr 9. PMID 18397542
- [Background] Witkowski JA, Parish LC. The assessment of acne: an evaluation of grading and lesion counting in the measurement of acne. Clin Dermatol. 2004 Sep-Oct;22(5):394-7. doi: 10.1016/j.clindermatol.2004.03.008. PMID 15556725